CLINICAL TRIAL: NCT05198388
Title: Beta Endorphins,Interleukin 1 and Interleukin 38 in Covid Patients Associated With Neuropsychological Manifestations.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, somaya redwan younes, Assistant Lecturer, Assiut University
Other Study IDs: covid study
Record Dates: First submitted 2022-01-19; First posted 2022-01-20 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Covid Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: βeta endorphins, interleukin 6 and interleukin 38 — * - Collection of peripheral blood samples in gel tube.
  * - Creparation of samples in centrifuge to obtain serum.
  * - Measurement of interleukin 6 and interleukin 38 and βeta endorphins using ELISA method.

SUMMARY:
Measurement of Beta endorphins,interleukin 1 and interleukin 38 in covid patients associated with neuropsychological manifestations.

DETAILED DESCRIPTION:
The world is facing one of its worst infectious disease pandemics in history, i.e., Covid-19. Coronavirus, SARS-CoV-2 was identified as the cause of an outbreak of a severe pneumonia-like disease, currently known as Covid-19. When COVID-19 infect the upper and lower respiratory tract it can cause mild or highly acute respiratory syndrome with consequent release of pro-inflammatory cytokines, including interleukin (IL)-1β and IL-6. (Herold T., et al., 2020) Although the main risks of COVID-19 is to cause injuries to the upper and lower respiratory track and lung, other organs are also affected including CNS leading to variety of neuropsychatric symptoms including headache, depression, and memory impairment.These psychological symptoms become more obvious by quarantine which is one of the most common protections against virus infections .These psychological symptoms also aasociated with alteration of level of beta endorphins. (Long B et al.,2020).

β-Endorphin, a morphine-like peptide, was identified in brain as an endogenous opioid peptide hormone that is produced and secreted in the pituitary gland and related to pain modulation and strongly linked to chronicity and severity of depression. The specific receptor for β-endorphin is the μ-opioid receptor. (Tanaka et al., 2003) β-Endorphin stimulates chemotaxis of monocytes, their differentiation into macrophages, and production of reactive oxygen species, interleukin (IL)-1β, IL-10, interferon-γ, and tumor necrosis factor-α in monocytes/macrophages. The μ-opioid receptor is upregulated by IL-1α and IL-1β. (Gein et al.,2016) The psychological disorders caused by Covid-19 have significant effects on the immune system, resulting in mast cell activation, increased generation of cytokines like IL-1, IL-37, IL-6, and C-reactive protein. Endorphin release therapy (ERT) can be very effective to reactivate thymus gland, increase production of NK cells and CD4+ cells and inhibit CD8+cells, prevent, and reduce inflammation in Covid-19 patients, thereby reducing many complications and associated deaths. (Ahmadpoor P et al ., 2020 ) IL-38 is the newest cytokine of the IL-1 family members, produced by several immune cells including B cells and macrophages. IL-38 is a suppressor cytokine which inhibits IL-1β and other pro-inflammatory IL-family members. IL-38 is a potential therapeutic cytokine which inhibits inflammation in viral infections including that caused by coronavirus-19, providing a new relevant strategy. (Gómez-Rial J et al.,2020)

ELIGIBILITY:
Inclusion Criteria: Patients had positive throat swab. Patients had chest finding on CT

Exclusion Criteria:

Other respiratory diseases

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sixity patients diagnosed with Covid-19 (30 patients with neurological manifestations and 30 patients without neurological manifestations) 30 healthy individuals as control group with matched age and sex.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
- Detection of βeta endorphins, interleukin 6 and interleukin 38 in serum of COVID-19 patients. | 3 years
  - Detection of βeta endorphins, interleukin 6 and interleukin 38 in serum of COVID-19 patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
- Collection of peripheral blood samples in gel tube.
  * - Creparation of samples in centrifuge to obtain serum.
  * - Measurement of interleukin 6 and interleukin 38 and βeta endorphins using ELISA method.